CLINICAL TRIAL: NCT00101478
Title: Partnership Programs to Reduce Cardiovascular Disparities - Baltimore Partnership
Brief Title: Improving Cardiovascular Treatment Approaches Among Minorities
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HP-00040555; U01HL079151 (NIH)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to improve cardiovascular disease (CVD) outcomes in racial and ethnic minorities. Specifically, the study will aim to improve provider and patient approaches to treatment of hypertension and diabetes, respectively.

DETAILED DESCRIPTION:
BACKGROUND:

While there has been great progress in reducing CVD morbidity and mortality in the U.S. over the past 40 years, some minority groups have not shared fully in this progress and continue to have lower life expectancy and higher CVD morbidity. On average, minorities have less access to medical care, receive less aggressive care and fewer diagnostic and therapeutic cardiac procedures, and adhere poorly to prescribed medical regimens. Thus, research to reduce health disparities by improving CVD outcomes in minorities offers potential for a substantial positive public heath impact. Academic medical centers and institutions capable of carrying out such research, however, often lack access to and the trust of minority patients. Minority patients often receive fragmented care because they lack access to regular medical care, present to emergency departments rather than primary care physicians for complications of an advanced chronic CVD condition, and are less likely to follow medical regimens. Minority communities often harbor distrust of clinical research. Minority patients report greater satisfaction when receiving care from minority providers and are reluctant to receive treatment outside their minority healthcare serving systems.

In general, minorities have high rates of hypertension, elevated cholesterol, cigarette smoking, obesity, metabolic syndrome, and diabetes, as well as other behavioral, environmental, and occupational risk factors for cardiovascular diseases, such as sleep problems. These are all elements that contribute to excess CVD morbidity and mortality. The causes of minority health disparities are complex and incompletely understood. Although evidence of genetic, biologic, and environmental factors is well documented, poor outcomes are also attributed to under-treatment. Such under-treatment may be due to limited access to health care or, in some cases, break-down of the medical system, or failure of the physician and/or patient to allow for optimal health care, even when access is not impaired. The complex interactions of behavior, socio-economic status (SES), culture, and ethnicity are important predictors of health outcomes and sources of health disparities. Despite efforts to elucidate genetic and environmental risk factors and to promote cardiovascular health in high-risk populations, trends in CVD outcomes suggest that CVD health disparities continue to widen.

The Partnerships Program to Reduce Cardiovascular Health Disparities involves collaboration between minority healthcare serving systems (MSSs) that lack a strong research program and research-intensive medical centers (RIMCs) that have a track record of NIH-supported research and patient care. Each Partnership Program will: a) design and carry out multiple interdisciplinary research projects that investigate complex biological, behavioral, and societal factors that contribute to CVD health disparities and facilitate clinical research within the MSS to improve CVD outcomes and reduce health disparities, and b) provide reciprocal educational and skills development programs so that investigators are able to conduct research aimed at reducing cardiovascular disparities, thereby enhancing research opportunities and enriching cultural sensitivity and cardiovascular research capabilities at both institutions.

The Request for Applications for Partnership Programs to Reduce Cardiovascular Disparities was released in September 2003. The awards were made in September 2004.

DESIGN NARRATIVE:

The collaborative partnership between the Bon Secours Baltimore Health System (BSBHS) and the University of Maryland Baltimore (UMB) seeks to improve provider and patient approaches to treatment of hypertension and diabetes, respectively. UMB also aims to modify physician-related barriers to minority enrollment in clinical trials, and BSBHS to improve patient adherence to treatment plans. Through didactic training, UMB aims to build a sustainable research program at BSBHS; through cultural sensitivity training, BSBHS expects to enhance the disparities program at UMB. The relative impact of physician and/or patient interventions for controlling hypertension and diabetes will be assessed. This will be a hypothesis-testing, prospective study, with an experimental 2 X 2 factorial design; it will be a four-arm randomized controlled trial. Outcomes will include adherence and improved knowledge/awareness of guidelines (of patients and their physicians), as well as patient clinical and quality of life measures. The study will be powered for the proportion of patients who attain the set goal. There will be a target enrollment of 800 patients (400 each for hypertension and diabetes), to afford 80% (up to 90%) power and allow for 25% attrition. Logistic regression will be used for the probability of reaching goal, multiple linear regression will be used for relative changes in mmHg (hypertension) and HbAlc (diabetes), and survival analysis will be used to model time to reach goal. Measurements will be taken of improved adherence of diabetes patients as a result of BSBHS actively identifying access barriers. Measurements will also be taken of changes in the willingness of patients to enroll in clinical trials as a result of physician-targeted education. The study seeks to demonstrate a best practice model, based on a collaborative partnership, and build a self-sustained research program at BSBHS and an enhanced cardiovascular disparities program at UMB. Community entities will have full access to resources at both institutions, which in turn will have access to invaluable input and support from community groups.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled hypertension or diabetes

Exclusion Criteria:

* Medical condition that would prevent treatment for hypertension at the University of Maryland
* Medical condition that would prevent treatment for diabetes at Bon Secours
* Uninsured

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study groups will be selected from primary and family health clinics, community, and patients of physicians participating in the study.
Sampling Method: Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Saunders, MD, Principal Investigator — University of Maryland, Baltimore; Reed Winston, MD, Principal Investigator — Bon Secours Hospital Baltimore; Fadia T. Shaya, PhD, MPH, Principal Investigator — Universitiy of Maryland Baltimore; Wallace R. Johnson, MD, Principal Investigator — Bon Secours Hospital Baltimore
Locations (2):
- United States (2):
  - University of Maryland Baltimore, Baltimore, Maryland
  - Bon Secours Hospital, Baltimore, Maryland